CLINICAL TRIAL: NCT03714711
Title: Patient Pain and Opioid Use Profile After Total Hip and Total Knee Arthroplasty
Brief Title: Pain Profile and Pain Medication Use After THA and TKA
Status: Withdrawn | Type: Observational
Why Stopped: PI decided to close due to current funding and future funding constraints on internal studies.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00100351
Record Dates: First submitted 2018-09-24; First posted 2018-10-22 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Pain, Postoperative
Keywords: total hip replacement; total knee replacement
MeSH Terms: conditions — Pain, Postoperative | interventions — Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total hip arthroplasty: Patient who are scheduled to undergo total hip replacement.
  Interventions: Procedure: total hip arthroplasty
- Total knee arthroplasty: Patient who are scheduled to undergo total knee replacement.
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total hip arthroplasty — Total hip replacement
  Groups: Total hip arthroplasty
Procedure: total knee arthroplasty — Total knee replacement
  Groups: Total knee arthroplasty

SUMMARY:
The over-prescription and overuse of opioid medications in the United States has recently been recognized as an epidemic. A new law in North Carolina (STOP Act) is aimed to limit opioid prescriptions following any surgical procedure including total hip (THA) and total knee arthroplasty (TKA). However, there is limited evidence regarding patient's pain and actual opioid consumption following THA and TKA that can be used by practitioners as guidance adapting to the new law. The purpose of this study is to investigate patient's pain and pain medication use in the perioperative period (0-6 weeks) following THA and TKA to establish a pain profile and thereby investigating risk factor for increased postoperative pain and opioid pain medication requirements. This study aims to stratify a predication model of postoperative pain and opioid medication requirement after THA and TKA to identify patients with a high propensity for pain, improve preoperative patient education on postoperative pain expectations, thereby helping practitioners implement new postoperative prescriptions limits for THA and TKA patient.

DETAILED DESCRIPTION:
Number of subjects: Patient undergoing THA and TKA will be enrolled in this prospective study. Patients older than 18 years of age, with cell phones capable of text messaging, and who agree to participate in this study will be included. Patients who have their primary residence in Missouri will be excluded from this study due to the lack of a state wide narcotic prescription database in Missouri. Up to 240 patients will be enrolled to reach a minimum of 200 participants (100 THA, 100 TKA patients) with complete data from pre to 1 year postoperatively.

Preoperative questionnaires: Patient will be required to complete a preoperative pain catastrophizing score, abrief pain inventory, EQ-5D, a hip disability and osteoarthritis outcome score (HOOS JR.) or knee injury and osteoarthritis outcome score (KOOS JR.) and aAbaseline pain level on a visual analog scale (0-10) will be recorded.

Preoperative pain medication assessment: Preoperative controlled substance use will be assessed using the patient's state residence Controlled Substance Reporting System. Patient socioeconomic status, prior history of pain medication use, and history of drug abuse will be recorded.

Patient preoperative pain sensitivity testing: Patients will then undergo pain algometer testing (FPK algometer, Wagner Instruments, Greenwich CT) to establish an objective baseline pain tolerance. There is no risk to the patient with algometer testing. Pressure algometer testing will be performed in a standard fashion. The probe is applied at a 90 degree angle to the skin at a constant rate of 10kPa/s to minimize the impact of the examiner's reaction time on recorded pain thresholds. The participant is instructed by the measurer to say "stop" when the sensation of pressure became the very first sensation of pain. There will be three spots to test patients, one for familiarity of the testing and the other 2 for data collection. This is initially performed once on ipsilateral the tibialis anterior as a "warm up." Then 3 measurements are taken on the operative medial epicondyle (for TKA) or ipsilateral lateral iliac crest (for THA) and averaged for the official score. Lastly, 3 measurements are also taken on the contralateral olecranon to measure systemic pain sensitivity. If the contralateral elbow has had prior surgery or active bursitis, the ipsilateral elbow will be used. Of important note, the algometer has a max force lock out of 100N to prevent any harm to the patient. In addition, we will capture dominant handgrip strength measured by the average of 3 attempts on a standard dynamometer.

In-hospital and postoperative pain and medication assessment: Patient's pain scores on an analog scale will be recorded daily from the patient's electronic medical record (lowest, highest, median) while admitted to the hospital. Patient will be contacted daily via text message to report pain scores and pain medication use. Text messaging via cell phones has become very common in the US and has been shown to be efficacious in obtaining longitudinal research data, specifically in assessing pain scores. Patient will be contacted daily via text messaging (Mosio, Seattle, WA).Mosio is a two-way mobile messaging platform that deploys automated text messages to study subjects. Subjects reply to the questions bv text message which are sent and received through mosio.

The participants will be asked the following questions by text messaging daily:

1. What was the average pain level (0-10) in the past 24 hours?
2. What was the highest level of satisfaction (0-10) with the total joint in the past 24 hours?
3. How many pain medication pills were taken in the past 24 hours?

The responses by the patient are replied to and typed as a standard text message. The answers will be captured by mosio and transferred in the secure database. The study team has instant access to the data server via secured log in authentication. Study replies can be downloaded as excel spreadsheets for further analysis.

At the standard of care 6-week and 1-year postoperative visit, participants will complete a Visual Analog Scale (VAS), PROMIS pain scale, EQ-5D and HOOS JR or KOOS JR questionnaire. Once questionnaires are completed this will conclude study participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age undergoing primary total hip or total knee replacement
* Able to give consent to participate in the study
* Patients have a cell phone capable of text messaging

Exclusion Criteria:

* Patients from states in the US without a narcotic prescription database (Missouri)
* Patients with previous joint surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary total hip or knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Pain level | 1 - 6 weeks on average
  Change in Patients' pain level on visual analog scale from 0-10; 0 no pain, 10 worst pain imaginable

SECONDARY OUTCOMES:
Change in opioid consumption | daily for 6 weeks after surgery
  Change in patient use of opioid pain medication
Change in satisfaction level | daily for 6 weeks after surgery
  Change in patient satisfaction with total joint replacement, scale 0-10; 0 no satisfaction, 10, highest satisfaction possible
EQ5D | Once before surgery, up to 10 minutes
  Health related quality of life; scale of 0-100, 0 worst health imaginable, 100 best health imaginable
EQ5D | 6 weeks postoperative
  Health related quality of life; scale of 0-100, 0 worst health imaginable, 100 best health imaginable
EQ5D | 1 year postoperative
  Health related quality of life; scale of 0-100, 0 worst health imaginable, 100 best health imaginable
hip disability and osteoarthritis outcome score (HOOS) | Once before surgery, up to 10 minutes
  Total hip replacement clinic outcome measure; scale from 0-100; 0 total hip disability, 100 perfect hip health
hip disability and osteoarthritis outcome score | 6 weeks postoperative
  Total hip replacement clinic outcome measure; scale from 0-100; 0 total hip disability, 100 perfect hip health
hip disability and osteoarthritis outcome score | 1 year postoperative
  Total hip replacement clinic outcome measure; scale from 0-100; 0 total hip disability, 100 perfect hip health
knee disability and osteoarthritis outcome score | Once before surgery, up to 10 minutes
  Total knee replacement clinic outcome measure; scale from 0-100; 0 total knee disability, 100 perfect knee health
knee disability and osteoarthritis outcome score | 6 weeks postoperative
  Total knee replacement clinic outcome measure; scale from 0-100; 0 total knee disability, 100 perfect knee health
knee disability and osteoarthritis outcome score | 1 year postoperative
  Total knee replacement clinic outcome measure; scale from 0-100; 0 total knee disability, 100 perfect knee health
Pain threshold | Preoperative clinic visit, up to 10 minutes
  Pressure algometer testing

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Seyler, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No